CLINICAL TRIAL: NCT05794958
Title: A Phase Ib, Open Label Study to Evaluate Safety of Axicabtagene Ciloleucel Reinfusion (Axi-Cel-2) in Patients With Relapsed and/or Refractory Second Line High-Risk Non-Hodgkin Lymphoma After Standard of Care Axi-Cel
Brief Title: Evaluate Safety of Axicabtagene Ciloleucel Reinfusion (Axi-Cel-2) in Patients With Relapsed and/or Refractory Second Line High-Risk Non-Hodgkin Lymphoma After Standard of Care Axi-Cel
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Kite Pharma (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB-68723; CCT5068 (Other: OnCore); NCI-2023-05593 (Registry Identifier: CTRP)
Record Dates: First submitted 2023-03-20; First posted 2023-04-03 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Non-Hodgkin Lymphoma; Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — axicabtagene ciloleucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Safety Run-in phase (Active Comparator): First three patients (maximum of 6) will receive 0.5 x 106/kg CART cells (25% standard dose) as reinfusion product between days 7 through 14 if CRS/ICANS has resolved to a grade 1 or less.
  Interventions: Drug: Axicabtagene Ciloleucel
- Phase 1b (Experimental): Up to 20 evaluable subjects will receive the target dose of AxiCel infusion to evaluate efficacy of Axi-Cel-2 in adults with high risk relapsed/refractory LBCL
  Interventions: Drug: Axicabtagene Ciloleucel

INTERVENTIONS:
Drug: Axicabtagene Ciloleucel — Subjects will receive a re-infusion of Axi-Cel (Axi-Cel-2) if signs and symptoms of cytokine release syndrome (CRS) and Immune Effector Cell Associated Neurotoxicity Syndrome (ICANS) are ≤ grade 1.
  Other Names: (Axi-cel-2)

SUMMARY:
This is a phase Ib study to establish safety of Axi-Cel-2 in patients with Large B Cell Lymphoma (LBCL) who are at high risk of relapse.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis: Histologically confirmed aggressive B cell NHL including the following types defined by WHO 2008:

   * Diffuse large B cell lymphoma (DLBCL); OR
   * primary mediastinal (thymic) large B cell lymphoma; OR
   * transformation of follicular lymphoma (TFL), marginal zone lymphoma to DLBCL; OR
   * high grade B-cell Lymphoma NOS will also be included
2. Patients must be considered high-risk lymphoma (defined as LDH greater than upper limit of normal per institutional cut-off) at or within two weeks of leukapheresis.
3. Subjects must have received at least and a maximum one prior line of therapy for LBCL indication (i.e subjects receiving second line standard of care Axi-Cel will be enrolled in this study).
4. At least 1 measurable lesion on PET-CT or CT scan. If the only measurable disease is lymph-node disease, at least 1 lymph node should be ≥ 1.5 cm.
5. Age 18 years or older
6. Eastern cooperative oncology group (ECOG) performance status of 0 or 1. ECOG 2 permitted if performance status is solely attributed to lymphoma.
7. Normal Organ and Marrow Function

   * ANC ≥ 1,000/uL
   * Platelet count ≥ 75,000/uL
   * Adequate renal, hepatic, pulmonary and cardiac function defined as:

     * Creatinine clearance (as estimated by Cockcroft Gault Equation) ≥ 60 mL/min
     * Serum ALT or AST ≤ 2.5 x ULN (except in subjects with liver involvement by lymphoma)
     * Total bilirubin ≤ 1.5 mg/dl, except in subjects with Gilbert's syndrome.
     * Cardiac ejection fraction ≥ 40%, no evidence of pericardial effusion as determined by an Echocardiogram.
   * No clinically significant pleural effusion or ascites
   * Baseline oxygen saturation > 92% on room air
8. Ability to understand and the willingness to sign the written IRB-approved informed consent document. Subjects unable to give informed consent will not be eligible for this study.
9. Females of childbearing potential must have a negative serum or urine pregnancy test (females who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential)
10. Contraception: Subjects of child-bearing or child-fathering potential must be willing to practice birth control from the time of enrollment on this study and for twelve (12) months after receiving the preparative lymphodepletion regimen.
11. If prior CD19 directed therapy, demonstrates CD19 positivity by biopsy (Flow cytometry or immunohistochemistry per the institutional criteria)
12. Prior therapy washout of at least 2 weeks or 5 half-lives, whichever is shorter, must have elapsed since any prior systemic therapy at the time the subject is planned for leukapheresis

Exclusion Criteria:

1. Prior treatment with CAR-T or adoptive cell therapy.
2. Prior allogeneic transplant.
3. No bridging therapy permitted except for steroids or radiotherapy (bridging therapy with steroids e.g. dexamethasone 40 mg for 5 days or radiotherapy is permitted). Measurable non-irradiated lesion post-apheresis needed for enrollment.
4. Active central nervous system disease from lymphoma. MRI of the brain with no evidence of CNS lymphoma if prior history of CNS involvement.
5. Prior history of allergic reactions or severe infusion reaction to Axi-Cel or any of the reagents used in the Axi-Cel infusion.
6. History of Richter's transformation of chronic leukemic lymphoma, small lymphocytic lymphoma, or lymphoplasmacytic lymphoma.
7. Any medical condition that in the judgement of the investigator is likely to interfere with assessment of safety or efficacy of study treatment.
8. Women who are pregnant or breastfeeding
9. History of invasive malignancy unless the patient has been disease-free for five years.

   * Exception: Nonmelanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, and breast) is eligible.
   * Hormonal therapy in subjects in remission >1 year will be allowed.
10. History of stroke or transient ischemic attack within 12 months before enrollment, or seizure disorders requiring active anticonvulsive medication.
11. In the investigator's judgment, the subject is unlikely to complete all study specific visits or procedures, including follow-up visits, or comply with the study requirements for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2038-04-01 (Estimated); Study Completion 2038-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of toxicities,dose limiting toxicity (DLT) of a second dose of AxiCel (Axi-Cel2) in adults with relapsed/refractory high-risk LBCL. | 28 days
  Subjects will be assessment for dose limiting toxicity (DLT) for 28 days after the infusion of Axi-Cel-2

SECONDARY OUTCOMES:
Progression free survival (PFS) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Saurabh Dahiya, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States